CLINICAL TRIAL: NCT04248114
Title: The Natural Neck Crease as an Anatomic Landmark for Thyroid Surgery Incision
Brief Title: Skin-crease Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Ronen Ohad, Director Head and Neck Unit, Western Galilee Hospital-Nahariya
Other Study IDs: NHR-014417
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound of the Neck — Anatomical measurements were performed on participants during an ultrasound exam

SUMMARY:
We performed a retrospective observational-analytic study. Anatomical measurements were performed on 118 participants during an ultrasound exam, and demographic data was collected from their medical files. The data was stratified according to age, sex, patient's body mass index (BMI), and height.

DETAILED DESCRIPTION:
Approval - Ethical Considerations The study was approved by the Institutional Review Board (NHR-014417). Study Design In this retrospective observational-analytic study we analyzed the anatomical relation between the cricoid cartilage, thyroid gland isthmus, and the superficial second neck crease. We reviewed patient data from between November 2016 and August 2018. The data was collected during ultrasound exams of 118 subjects who underwent assessment of the thyroid gland. Patients who had any neck surgical procedure prior to the test, patients with abnormalities in the anterior neck, and patients without clear second crease were excluded.

During the examination, patients were lying supine with their head in mild extension, in the same manner that is practiced during a thyroidectomy. The assessment and collection of data was performed by the senior author (OR) who routinely performs both this preoperative examination and thyroid surgeries in the medical center. The precise location of the cricoid cartilage and the thyroid isthmus was determined using ultrasound. The main parameters were the distances between the thyroid isthmus superior border and the second neck crease, and the distance between the cricoid cartilage superior border and the second neck crease. These were measured with a ruler with ultrasound imaging guidance (Figure 1).

Several neck creases can be observed in normal adults. The first upper crease runs horizontally roughly along the thyroid notch and hyoid bone. A second lower neck crease runs parallel to it approximately at the height of the cricoid and this is the crease the measurements in our study relate to. Occasionally there is a third prominent skin crease around 2-3 finger breadths above the clavicle. Other less prominent horizontal neck creases can be present.

Demographic variables, such as age, sex, BMI, and height, were collected from medical records and used for result stratification either as continuous variables or divided into sub-groups according to accepted divisions.

Sample size calculation The hypothesis was that the second neck crease is superficial to the thyroid gland isthmus superior border (0 cm horizontal distance). A vertical distance of 0.5 cm and more was considered significant difference in the location.

Statistical analysis Distance between the thyroid isthmus or the cricoid cartilage and the second neck crease were described by means, standard deviation, and range. Age, sex, BMI, and height were analyzed as quantitative variables with the measures mentioned above. The continuous variants were also grouped for a clearer presentation of the results. The BMI variant was categorized into accepted ranges: underweight (below 18.5 kg/m2), normal weight (18.5 to 25 kg/m2), overweight (25 to 30 kg/m2), and obese (over 30 kg/m2). BMI sub-groups and sex variables were described by frequencies and percentages.

The distances were compared among sub-groups using ANOVA, Kruskal-Wallis test, Independent sample t-test, and Wilcoxon rank sum test. The choice between those tests was according to the number of sub-groups, the group's sample size, and the distribution of the data in each sub-group.

A correlation between age, BMI, height, and the distance was tested by Pearson's correlation coefficient test or Spearman's correlation coefficient test. The choice between those tests was according to the sample size and the score's distribution. If the variable was defined as ordinal sub-groups, Spearman's correlation coefficient test was used.

ELIGIBILITY:
Inclusion Criteria:

Subjects who underwent assessment of the thyroid gland

Exclusion Criteria:

Patients who had any neck surgical procedure prior to the test, patients with abnormalities in the anterior neck, and patients without clear second crease were excluded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data was collected during ultrasound exams of subjects who underwent assessment of the thyroid gland.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
anatomical relations between the second neck skin crease and the thyroid gland isthmus and cricoid cartilage | June 1st 2016 until August 31 2018
  Several neck creases can be observed in normal adults. The first upper crease runs horizontally roughly along the thyroid notch and hyoid bone. A second lower neck crease runs parallel to it approximately at the height of the cricoid; the measurements, in centimeters, in our study relate to this crease.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fancy T, Gallagher D 3rd, Hornig JD. Surgical anatomy of the thyroid and parathyroid glands. Otolaryngol Clin North Am. 2010 Apr;43(2):221-7, vii. doi: 10.1016/j.otc.2010.01.001. PMID 20510710
- [Result] Brunaud L, Zarnegar R, Wada N, Ituarte P, Clark OH, Duh QY. Incision length for standard thyroidectomy and parathyroidectomy: when is it minimally invasive? Arch Surg. 2003 Oct;138(10):1140-3. doi: 10.1001/archsurg.138.10.1140. PMID 14557134
- [Result] Choi Y, Lee JH, Kim YH, Lee YS, Chang HS, Park CS, Roh MR. Impact of postthyroidectomy scar on the quality of life of thyroid cancer patients. Ann Dermatol. 2014 Dec;26(6):693-9. doi: 10.5021/ad.2014.26.6.693. Epub 2014 Nov 26. PMID 25473220